CLINICAL TRIAL: NCT00237614
Title: Contrast Nephropathy Prevention With N-Acetylcysteine in Acute Myocardial Infarction
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: University of Milan (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: CCS16 RC/2003
Record Dates: First submitted 2005-10-07; First posted 2005-10-12 (Estimated); Last update posted 2006-07-18 (Estimated); Status verified 2005-07

CONDITIONS: Contrast-Induced Nephropathy; Acute Myocardial Infarction
Keywords: Contrast-induced nephropathy; Acute myocardial infarction; Primary coronary angioplasty
MeSH Terms: interventions — Acetylcysteine

INTERVENTIONS:
Drug: intravenous and oral N-acetylcysteine

SUMMARY:
Patients with acute myocardial infarction undergoing primary angioplasty are at high risk for renal injury due to the toxic effect of contrast agents. Patients developing renal dysfunction after primary angioplasty have worse outcome. To investigate the role of the antioxidant N-acetylcysteine (NAC) in preventing renal injury in angioplasty, we randomized 352 consecutive patients undergoing primary angioplasty into three groups: the first group received NAC at standard dose (NAC group, 600 mg i.v. bolus before primary angioplasty, followed by oral 600 mg twice daily for the following 48 hours; n=115), the second group received NAC at double dose (DD-NAC group; 1,200 mg i.v. bolus and oral 1,200 mg twice daily for 48 hours; n=118), and the last group received placebo (controls; n=119).

ELIGIBILITY:
Inclusion Criteria:Consecutive patients admitted to the Coronary Care Unit for ST-segment elevation acute myocardial infarction undergoing primary angioplasty. Patients were included if they presented within 12 hours (18 hours for acute myocardial infarction complicated by cardiogenic shock) from the onset of symptoms. -

Exclusion Criteria:Patients in chronic peritoneal or hemodialytic treatment and those with known allergy to N-acetylcysteine.

-

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300
Dates: Start 2003-02; Study Completion 2005-05

PRIMARY OUTCOMES:
Incidence of contrast-induced nephropathy

SECONDARY OUTCOMES:
In-hospital major clinical adverse events including death

CONTACTS AND LOCATIONS:
Overall Officials: Antonio L Bartorelli, MD, Study Director — Centro Cardiologico Monzino
Locations (1):
- Centro Cardiologico Monzino, Milan, Italy

REFERENCES:
- [Background] Marenzi G, Lauri G, Assanelli E, Campodonico J, De Metrio M, Marana I, Grazi M, Veglia F, Bartorelli AL. Contrast-induced nephropathy in patients undergoing primary angioplasty for acute myocardial infarction. J Am Coll Cardiol. 2004 Nov 2;44(9):1780-5. doi: 10.1016/j.jacc.2004.07.043. PMID 15519007
- [Result] Marenzi G, Assanelli E, Marana I, Lauri G, Campodonico J, Grazi M, De Metrio M, Galli S, Fabbiocchi F, Montorsi P, Veglia F, Bartorelli AL. N-acetylcysteine and contrast-induced nephropathy in primary angioplasty. N Engl J Med. 2006 Jun 29;354(26):2773-82. doi: 10.1056/NEJMoa054209. PMID 16807414